CLINICAL TRIAL: NCT03097822
Title: Response Prediction After Gamma Knife Surgery (GKS) in Patients With Vestibular Schwannoma Using Dynamic Contrast-Enhanced (DCE) MR Imaging
Brief Title: Response Prediction After GKS in Patients With Vestibular Schwannoma Using DCE MR Imaging
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Seung Hong Choi, SeoulNUH, Seoul National University Hospital
Other Study IDs: H-1611-087-809
Record Dates: First submitted 2017-03-20; First posted 2017-03-31 (Actual); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Vestibular Schwannoma
MeSH Terms: conditions — Neuroma, Acoustic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Response Prediction after Gamma Knife Surgery (GKS) in Patients with Vestibular Schwannoma using Dynamic Contrast-Enhanced (DCE) MR Imaging

DETAILED DESCRIPTION:
The purpose of this study was to evaluate the response of Gamma Knife Surgery to Ktrans, Ve, and Vp, which are indicators of permeability map obtained from dynamic contrast enhanced (DCE) MRI in patients with vestibular schwannoma .

ELIGIBILITY:
Inclusion Criteria:

* Patients with vestibular schwannoma, who underwent gamma knife surgery and pre-op dynamic contrast enhanced (DCE) MRI
* Patients with vestibular schwannoma, who received consent

Exclusion Criteria:

* In addition to the vestibular schwannoma, if the brain has other underlying or systemic disease
* During the observation period, other treatments were performed other than gamma knife surgery
* If patients have a contraindication to MRI (eg, pacemaker, cochlear implants, hemodynamically unstable)
* Concomitant use of gadolinium MRI contrast agents (eg, renal insufficiency [glomerular filtration rate <30 ML / min]), or if there was a side effect when using a contrast medium.
* Adults with impaired ability to cope
* If the images and medical records required for this study are not available or are not appropriate

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with vestibular schwannoma, who underwent gamma knife surgery
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Tumor size change before and after surgery | pre-op, Immediately after surgery

SECONDARY OUTCOMES:
In patients who underwent gamma knife surgery, the magnitude of tumor size change before and after surgery | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: SeungHong Choi, MD,PhD, Principal Investigator — Seoul National University Hospital(Radiology)